CLINICAL TRIAL: NCT07128758
Title: The Effect of Music Listening on the Initial Mobility Level of Pediatric Patients Undergoing Appendectomy: A Randomized Controlled Trial
Brief Title: Effect of Music Listening on Early Mobility in Children Undergoing Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma Dilek Turan, Assoc. Prof., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FDilekTuran
Record Dates: First submitted 2025-07-30; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Appendectomy; Child; Mobility; Mobilization; Music Listening Intervention
Keywords: Appendectomy; Child; Initial Mobility; Mobilization; Music Listening

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group Implementation (Experimental): Before surgery, children were asked whether they enjoyed listening to music and what styles of music they liked.
  * A 30-minute playlist was created using songs from the music pool based on the child's preferences.
  * Children were informed about postoperative mobility and which movements they would be expected to perform.
  Interventions: Behavioral: Music Group Implementation Before surgery, children were asked whether they enjoyed listening to music and what styles of music they liked.
- Control Group (No Intervention): No music Listening

INTERVENTIONS:
Behavioral: Music Group Implementation Before surgery, children were asked whether they enjoyed listening to music and what styles of music they liked. — All procedures required for developing a music pool to be used for music listening intervention in children undergoing appendectomy were completed and are outlined as follows:
  * Children were asked about their music preferences.
  * Songs were selected from the Ministry of National Education's music books.
  * Music with proven effectiveness was selected from music platforms.
  * A music pool was created by the researcher based on these inputs.
  * Expert opinions were obtained from 12 academicians and 10 healthy children regarding the music pool.
  * Necessary revisions were made in line with expert feedback, and the final version of the music pool was determined.
  * A pilot application was conducted (data from the pilot were not included in the main data set).
  * Children were randomly assigned to the music and control groups using randomization (https://www.random.org).
  * A neutral observer (not the researcher/a blinded observer) was trained to administer the scales after the music intervention
  Arms: Music Group Implementation

SUMMARY:
This randomized controlled study aimed to evaluate the effect of music listening on the initial mobility level of children who underwent appendectomy. The study was conducted at Ankara Etlik City Hospital, Pediatric Surgery Clinic, between March and May 2025. A total of 68 children aged 6-18 years, with no other systematic diseases and who consented to participate, were included. The music group consisted of 34 children and the control group of 34. A specially designed music pool, tailored separately for 6-11 and 12-18 age groups, was developed through child interviews, expert opinions, national education materials, and evidence-based motivational music. Children in the music group listened to music postoperatively, while the control group received only standard clinical care. Data were collected using the Child Information Form, Patient Mobility Scale, and Observer Mobility Scale.

ELIGIBILITY:
Inclusion Criteria:

* The child must have undergone an appendectomy.
* Be between the ages of 6 and 18.
* Have no motor impairments that would impede mobility.
* Have no additional chronic/systemic diseases.

Exclusion Criteria:

* Refusal to continue participating in the study at any stage.
* Refusal to participate in the first mobility measurement of the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Patient Mobility Score (Patient Mobility Scale Score) | immediately after the surgery
  Completed by the patient. The six-item scale evaluates three key postoperative mobilization activities: sitting on the bedside, standing at the bedside, and walking in the patient room. Each item is scored between 0 and 15, with the total scale score ranging from 0 to 90. Higher scores indicate greater pain and difficulty during mobilization, while lower scores reflect reduced pain and ease of movement.
The Observer Mobility Score (The Observer Mobility Scale Score) | immediately after the surgery
  Completed by the observer. The Observer Mobility Scale developed by the same authors as a complementary dimension to the Patient Mobility Scale, evaluates objective observations of the same three postoperative activities. Each item is scored on a scale of 1 to 5, with a total score range of 3 to 15. Higher scores reflect poorer mobility performance, while lower scores indicate better and more adequate postoperative mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Dilek Turan, PhD, Study Director — Akdeniz University; Özgür Çağlar, MD, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The article is considered to be shared after it is accepted in a journal and published.

REFERENCES:
- [Background] Islam T, Sagor MS, Tamanna NT, Bappy MKI, Danishuddin, Haque MA, Lackner M. Exploring the Immunological Role of the Microbial Composition of the Appendix and the Associated Risks of Appendectomies. J Pers Med. 2025 Mar 14;15(3):112. doi: 10.3390/jpm15030112. PMID 40137428
- [Background] Pratiwi, E. and F.M. Said, The role of paediatric nurse to enhance atraumatic care for hospitalised children: Literature review. Malaysian Journal of Medical Research, 2025. 9(1): p. 42-51.
- [Background] Prastyo, W.A. and A.I. Nugraheni, Management strategies and surgical outcomes for pediatric appendicitis: A literature review. The Indonesian Journal of General Medicine, 2025. 10(2): p. 11-24.
- [Background] Selvaggi L, Pata F, Pellino G, Podda M, Di Saverio S, De Luca GM, Sperlongano P, Selvaggi F, Nardo B. Acute appendicitis and its treatment: a historical overview. Int J Colorectal Dis. 2025 Jan 30;40(1):28. doi: 10.1007/s00384-024-04793-7. PMID 39881071